CLINICAL TRIAL: NCT06636383
Title: GSDIa Disease Monitoring Program
Brief Title: Glycogen Storage Disease Type Ia (GSDIa) Disease Monitoring Program
Status: Recruiting | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DTX401-CL401; 2023-510219-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-20; First posted 2024-10-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glycogen Storage Disease Type Ia
Keywords: Glycogen storage disorder Ia; AAV; Gene therapy; Von Gierke disease; Glucose metabolism disorder; GSD1; GSDIa
MeSH Terms: conditions — Hepatorenal form of glycogen storage disease; Glycogen Storage Disease Type I; Glucose Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: DTX401 in Prior Clinical Study: Patients administered DTX401(pariglasgene brecaparvovec), full or partial dose, in prior clinical study involving DTX401
  Interventions: Other: No Intervention
- Group 2: DTX401 in Post-Marketing Setting: Patients administered prescribed DTX401(pariglasgene brecaparvovec), full or partial dose, in a post-marketing setting
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No investigational/study product will be administered in this DMP.

SUMMARY:
The main objective of this observational study is to evaluate the long-term safety and effectiveness of DTX401 for at least 10 years after DTX401 administration.

DETAILED DESCRIPTION:
The DTX401-CL401 Disease Monitoring Program (DMP) is a prospective, multicenter, long-term observational study to follow up participants with GSDIa for at least 10 years after the administration of DTX401.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had:

  * DTX401 (full or partial dose) administered in a parent clinical study (Group 1) or
  * Prescribed DTX401(full or partial dose) administered in a post-marketing setting (Group 2)
* Patient is willing and able to provide informed consent after the nature of the study has been explained, and prior to any research-related assessments or procedures. If a minor or an adult with cognitive limitations, the patient is willing and able (if possible) to provide assent and have a legally authorized representative provide informed consent after the nature of the study has been explained, and prior to any research-related assessments or procedures.

Exclusion Criteria:

* Presence of any condition that would interfere with study participation, interpretation of results or affect patient's safety in the opinion of the Investigator

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who received DTX401 in a qualifying clinical study will be expected and asked to participate in the DMP upon completion or early termination (ET) from the parent study, as required by regulatory agencies for all gene therapy studies.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2036-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Serious Adverse Events (SAEs) Assessed as Related to DTX401 by the Investigator | 10 Years
Incidence, Relationship, Severity and Seriousness of Adverse Events of Special Interest (AESIs) for Adeno-Associated Virus (AAV) Therapies | 10 Years
Incidence of Pregnancy in Patients Treated with DTX401 or Patient's Partner | 10 Years
Outcomes of Pregnancy in Patients Treated with DTX401 or Patient's Partner | 10 Years
Incidence and Severity of SAEs of Infusion-Related Reactions Including Hypersensitivity (Group 2 only) | 1 Year
Incidence and Severity of SAEs Assessed by the Investigator as Related to Concomitant Immunomodulatory Therapies (Group 2 only) | 1 Year

SECONDARY OUTCOMES:
Percent Change Over Time from Baseline in Total Cornstarch Intake | Baseline, Up to 10 Years
Change from Baseline Over Time in Frequency of Cornstarch Intake | Baseline, Up to 10 Years
Change from Baseline Over Time in Number of Nighttime Awakenings for Cornstarch | Baseline, Up to 10 Years
Change from Baseline Over Time in Dependance on Continuous Overnight Tube Feeding for Exogenous Glucose Delivery | Baseline, Up to 10 Years
Change from Baseline Over Time in Daily Dietary Intake of Foods, Beverages, and Medical Foods/Formulas (Non-Cornstarch) | Baseline, Up to 10 Years
Change from Baseline Over Time in Daytime and Nighttime Percentage of Glucose Values During the 2 Weeks Leading Up to the Assessment Visits | Baseline, Up to 10 Years
  The following ranges will be assessed: < 54 mg/dL, < 60 mg/dL, < 70 mg/dL, 70-120 mg/dL, > 120 mg/dL
Change from Baseline Over Time in Total Number of Hypoglycemic Events on Continuous Glucose Monitoring (CGM) During the 2 Weeks Leading Up to the Assessment Visits | Baseline, Up to 10 Years
  The following ranges will be assessed: < 54 mg/dL, < 70 mg/dL
Change from Baseline Over Time in Total Duration of Hypoglycemic Events on CGM During the 2 Weeks Leading Up to the Assessment Visits | Baseline, Up to 10 Years
  The following ranges will be assessed: < 54 mg/dL, < 70 mg/dL
Change from Baseline Over Time in Real-World Overnight Fasting Tolerance | Baseline, Up to 10 Years
Change from Baseline Over Time in Metabolic and GSDIa Related Parameters: Height | 10 Years
Change from Baseline Over Time in Metabolic and GSDIa Related Parameters: Weight | 10 Years
Change from Baseline Over Time in Metabolic and GSDIa Related Parameters: Body Mass Index (BMI) | 10 Years
Number of Participants with Clinically Significant Laboratory Values | 10 Years
Frequency of Major Clinical Events (MCEs) | 10 Years
Frequency of MCEs from Review of Medical Records | 10 Years
Change from Baseline in Patient Experience Clinical Interview | Baseline, Up to 10 Years
Change from Baseline in European Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) Questionnaire Score | Baseline, Up to 1 Year
Change from Baseline in European Quality of Life 5 Dimensions Youth (EQ-5D-Y) Questionnaire Score | Baseline, Up to 1 Year
Change from Baseline Over Time in Annual Number of GSDIa Related Hospitalizations, Emergency Room Visits, Outpatient Visits, and Hospital Days | Baseline, Up to 10 Years
Change from Baseline Over Time in Missed Work/School Days in the Past 3 Months | Baseline, Up to 10 Years
Change from Baseline in Work/School Productivity Rating | Baseline, Up to 10 Years
Change from Baseline in Employment | Baseline, Up to 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceuticals Inc.
Locations (19):
- United States (9):
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Denver, Colorado
  - University of Connecticut Health Center, Hartford, Connecticut
  - University of Michigan, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul, Brazil
- McGill University Health Center, Montreal, Quebec, Canada
- Rigshospitalet, Copenhagen, Denmark
- Universitätsklinikum Hamburg Eppendorf, Hamburg, Germany
- Italy (2):
  - University of Naples, Napoli, Campania
  - Istituto G Gaslini Ospedale Pediatrico IRCCS, Genoa
- Japan (2):
  - Osaka City General Hospital, Osaka
  - Fujita Health University Hospital, Toyoake
- Groningen University, Groningen, Provincie Groningen, Netherlands
- Hospital Clínico Universitario de Santiago, Santiago, Spain

REFERENCES:
- See also: Our Clinical Trial Transparency Commitment-Ultragenyx — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/
- See also: Ultragenyx Patient Advocacy Website — https://www.ultrarareadvocacy.com/conditions-we-study/glycogen-storage-disease-type-ia-gsdia/